CLINICAL TRIAL: NCT06908551
Title: Pylorus Distensibility Measurement in Overweight and Obese (BMI 27-40) Patients
Brief Title: Pylorus Distensibility Measurement
Status: Not yet recruiting | Type: Observational
Sponsor: BariaTek Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-006-001
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims at characterizing the pylorus functionality in overweight and obese patients (BMI 27-40) using a systematic measurement approach by using an impedance planimetry technology.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 20 and 60 years inclusive
2. A BMI between 27.0 and 40.0 kg/m2
3. Willing and able to provide written informed consent
4. Willing and able to comply with the study procedures

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Overweight and obese (BMI 27-40)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Calculation of pylorus Cross Sectional Area | Baseline